CLINICAL TRIAL: NCT02042976
Title: A Randomised Controlled Trial of Mindfulness-based Cognitive Therapy (MBCT) for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Mindfulness-based Cognitive Therapy for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MBCT-KOL-2014
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Chronic Obstructive Lung Disease; Chronic Obstructive Airway Disease; Chronic Bronchitis; Emphysema
Keywords: Chronic obstructive pulmonary disease (COPD); Mindfulness-based cognitive therapy (MBCT); Behavioural intervention; Quality-of-life; Anxiety; Depression; Physical health status
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Anxiety Disorders; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based cognitive therapy + pulmonary rehabilitation (Experimental): An 8-week manual-based programme developed by Segal, Williams and Teasdale (2013) adjusted to the COPD population. The programme is delivered as an add-on to an 8-week standardised rehabilitation programme consisting of physical exercise and COPD-specific patient education.
  Interventions: Behavioral: Mindfulness-based cognitive therapy; Behavioral: Pulmonary rehabilitation
- Pulmonary rehabilitation only (Active Comparator): An 8-week standardised rehabilitation programme consisting of physical exercise and COPD-specific patient education.
  Interventions: Behavioral: Pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy
  Arms: Mindfulness-based cognitive therapy + pulmonary rehabilitation
Behavioral: Pulmonary rehabilitation

SUMMARY:
The purpose of the study is to determine the efficacy of mindfulness-based cognitive therapy (MBCT) as an add-on to pulmonary rehabilitation (treatment as usual, TAU) in chronic obstructive pulmonary disease (COPD).

The investigators hypothesize that compared to treatment-as-usual, the add-on of MBCT will result in improved psychological (anxiety, depression) and physical outcomes (physical health status, activity level, inflammatory markers). Furthermore, the investigators will explore the possible moderating role of individual differences in sociodemographic and disease-related characteristics and the perceived quality of the therapeutic alliance, as well as the mediating role of mindfulness, breathlessness catastrophizing, self-efficacy, and self-compassion for the hypothesised effect.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major burden for the affected patients, who are continuously struggling with the hallmark symptoms breathlessness, cough, and sputum together with high levels of anxiety and depression and impairment of quality of life (QoL). The potential value of complementary interventions in COPD has long been recognised, yet so far, no overall significant effects of psychosocial intervention programs such as cognitive behavioural therapy or supportive/analytical psychotherapy have been found.

Mindfulness-based interventions have been shown to improve levels of physical symptoms, stress, anxiety, depression, and QoL in other chronic conditions, and could also be relevant in COPD. The present randomized controlled trial will test the efficacy of mindfulness-based cognitive therapy (MBCT) in COPD patients. The investigators hypothesize that compared to treatment-as-usual, the add-on of MBCT will result in improved psychological (anxiety, depression) and physical outcomes (physical health status, activity level, inflammatory markers). Furthermore, the investigators will explore the possible moderating role of individual differences in sociodemographic and disease-related characteristics and the perceived quality of the therapeutic alliance, as well as the mediating role of mindfulness, breathlessness catastrophizing, self-efficacy, and self-compassion for the hypothesised effect.

Patients recruited from the Department of Respiratory Medicine, Aarhus University Hospital, will be randomized to participate in either an 8-week MBCT program as an add-on to the already established pulmonary rehabilitation program (intervention group) or pulmonary rehabilitation only (treatment-as-usual). Questionnaires assessing outcomes, mediators and moderators will be completed before, during, and after the intervention as well as at a 3 and 6 mo. follow-up.

This study will be one of the first to test the efficacy of MBCT in COPD, bringing attention to a patient group that is relatively ignored by the public as well as in the health psychological empirical literature.

After data collection, but prior to analysis, inaccuracies in the content of the registration were discovered. Some changes made prior to recruitment of the first participant had not been registered. The inaccuracies were amended in an update, 15 February 2017: 1) The primary outcome measure of iBODE (objective physical health status) was omitted (no data were collected). 2) The time frame for primary outcomes was changed from "Baseline, week 8" to "Baseline, 6 mo. follow-up". 3) Prior to data collection, three variables to be included in moderator and mediator analyses were added (therapeutic working alliance, mindfulness, and breathlessness catastrophizing).

ELIGIBILITY:
Inclusion Criteria:

* severe to very severe COPD
* motivated to participate in pulmonary rehabilitation
* sufficient mobility to attend pulmonary rehabilitation

Exclusion Criteria:

* certain comorbidities (e.g. unstable coronary complications, psychiatric illness)
* severe cognitive disability (e.g. dementia)
* inability to speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical health status impairment on the COPD Assessment Test (CAT) six months after termination of the 8-week treatment program | Baseline, 6-mo. follow-up
Change from baseline in anxiety and depression on the Hospital Anxiety and Depression Scale (HADS) six months after termination of the 8-week treatment program | Baseline, 6-mo. follow-up

SECONDARY OUTCOMES:
Change from baseline in physical activity at week 8 | Baseline, Week 8
  Measured by accelerometry
Change from baseline in inflammation at week 8 | Baseline, Week 8
  Measured by analysis of pro-inflammatory mRNA levels (IL-6, IL-8, IL-17E, TNF-alpha)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, MSc DMSci, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Background] Baraniak A, Sheffield D. The efficacy of psychologically based interventions to improve anxiety, depression and quality of life in COPD: a systematic review and meta-analysis. Patient Educ Couns. 2011 Apr;83(1):29-36. doi: 10.1016/j.pec.2010.04.010. Epub 2010 May 5. PMID 20447795
- [Background] Coventry PA, Gellatly JL. Improving outcomes for COPD patients with mild-to-moderate anxiety and depression: a systematic review of cognitive behavioural therapy. Br J Health Psychol. 2008 Sep;13(Pt 3):381-400. doi: 10.1348/135910707X203723. Epub 2007 Apr 18. PMID 17535503
- [Background] Rose C, Wallace L, Dickson R, Ayres J, Lehman R, Searle Y, Burge PS. The most effective psychologically-based treatments to reduce anxiety and panic in patients with chronic obstructive pulmonary disease (COPD): a systematic review. Patient Educ Couns. 2002 Aug;47(4):311-8. doi: 10.1016/s0738-3991(02)00004-6. PMID 12135822
- [Derived] Farver-Vestergaard I, O'Toole MS, O'Connor M, Lokke A, Bendstrup E, Basdeo SA, Cox DJ, Dunne PJ, Ruggeri K, Early F, Zachariae R. Mindfulness-based cognitive therapy in COPD: a cluster randomised controlled trial. Eur Respir J. 2018 Jan 31;51(2):1702082. doi: 10.1183/13993003.02082-2017. Print 2018 Feb. PMID 29386337